CLINICAL TRIAL: NCT05591781
Title: Efficacy of High Frequency Chest Wall Oscillations Versus Lung Flute in Chronic Obstructive Pulmonary Disease Postcovid
Brief Title: High Frequency Chest Wall Oscillations Versus Lung Flute in Chronic Obstructive Pulmonary Disease Post(SARS-CoV-2)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed El-Moatasem Mohamed, lecturer of physical therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003822
Record Dates: First submitted 2022-10-14; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Chest Wall Oscillation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Vest Airway Clearance System (Experimental): Thirty patients (Group A) received high frequency chest wall oscillation with vest system in addition to their prescribed medication, 3 times per week for three successive weeks and the total duration of each session was 15-30 minutes
  Interventions: Device: high frequency chest wall oscillation with vest system
- Lung flute (OPEP) (Active Comparator): Thirty patients (Group B) received Lung flute (OPEP) in addition to their prescribed medication, 3 times per week twice a day
  Interventions: Device: Lung flute (OPEP)

INTERVENTIONS:
Device: high frequency chest wall oscillation with vest system — Patients were assigned to 2 groups with pre- and post- treatment protocol application. All patients were thoroughly evaluated before and after treatment protocol application.
  Arms: Vest Airway Clearance System
Device: Lung flute (OPEP) — . Thirty patients (Group B) received Lung flute (OPEP) in addition to their prescribed medication, 3 times per week twice a day for three successive weeks
  Arms: Lung flute (OPEP)

SUMMARY:
COPD causes an acute deterioration of respiratory symptoms, particularly increased breathlessness and cough, and increased sputum volume and/or purulence. Worsening airflow limitation is associated with an increasing prevalence of exacerbations and risk of death. These exacerbations can range from self-limited diseases to episodes of florid respiratory failure requiring mechanical ventilation .Hospitalization for COPD patients post COVID is associated with poor prognosis with increased risk of death. Hence techniques of efficient clearance of peripheral airways may reduce airway occlusion by excess mucus and inflammatory cells, improving lung function, exercise capacity and reducing exacerbation frequency.

DETAILED DESCRIPTION:
Patients were assigned to 2 groups with pre- and post- treatment protocol application. All patients were thoroughly evaluated before and after treatment protocol application. Thirty patients (Group A) received high frequency chest wall oscillation with vest system in addition to their prescribed medication, 3 times per week for three successive weeks and the total duration of each session was 15-30 minutes. Thirty patients (Group B) received Lung flute (OPEP) in addition to their prescribed medication, 2 times per week twice a day for three successive weeks and the total duration of each session was 10-15 minutes

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 40-60 years old
* All patients were recovered from COVID not more than 3 months
* All patients were diagnosed as COPD for at least two years ago.
* All patients had irreversible/ partially reversible obstruction of airflow.
* COPD patients had a post-bronchodilator, FEV1/FVC% < 70%. They had an increase in FEV1< 200 ml, or < 12% of baseline value 20 minutes after 2 puffs of inhaled salbutamol (100 µg) given via a metered-dose inhaler.

Exclusion Criteria:

* Presence of malignant disease.

  * Patients with acute infection.
  * History of osteoporosis, significant gastro-oesophageal reflux, hiatus hernia.
  * Recent acute cardiac event (6 weeks) or congestive cardiac failure.
  * Any significant musculoskeletal disorders.

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | Forced vital capacity (FVC)will be measured at baseline, and after three weeks.
  FVC is the amount of air that can be forcibly exhaled from lungs after deepest inspiration, it's measured by spirometry
Forced expiratory volume in one second (FEV1) | FEV1 will be measured at baseline, and after three weeks.
  FEV1 is the maximum amount of air that the subject can forcibly expel during the first second following maximal inhalation
FEV1/FVC ratio | FEV1/FVC ratio will be measured at baseline, and after three weeks.
  The FEV1/FVC is a ratio that reflects the amount of air you can forcefully exhale from your lungs. It's measured by spirometry, a test used to evaluate lung function
The forced mid-expiratory flow (FEF25-75%) | (FEF25-75%) will be measured at baseline, and after three weeks.
  (FEF25-75) measures the average flow rates of medium-to-small airways during the forced vital capacity (FVC).it' is a potentially sensitive marker of obstructive peripheral airflow

SECONDARY OUTCOMES:
Six-minute walk test | 6min walk test will be measured at baseline, and after three weeks.
  Six-minute walk test was carried out before and after interventions to determine the patient functional capacity
COPD assessment test (CAT | COPD assessment test (CAT)will be measured at baseline, and after three weeks.
  is a validated, short (8-item) and simple patient completed questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt